CLINICAL TRIAL: NCT03819491
Title: Bioavailability Study of COQUN ORAL FORMULATION (CoQ10) Administered in Healthy Adults (CoQ10-01)
Brief Title: Bioavailability Study of COQUN ORAL FORMULATION
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VF-BAQ10/2018
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Male & Female Healthy Volunteers
Keywords: COQUN; antioxidant; Bioavailability; CoQ10; Healthy

STUDY DESIGN:
Intervention Model Description: To evaluate the best dosage between 100 mg OD or 100 mg BID for COQUN ORAL FORMULATION in order to reach a level of plasma concentration which might assure its antioxidant effect if taken on a regular basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 100 mg OD
  Interventions: Dietary Supplement: COQUN ORAL FORMULATION
- Group B (Experimental): 100 mg BID
  Interventions: Dietary Supplement: COQUN ORAL FORMULATION

INTERVENTIONS:
Dietary Supplement: COQUN ORAL FORMULATION — COQUN ORAL FORMULATION is a food supplement based on Coenzyme Q10 MINIACTIVES®

SUMMARY:
The goal of the study is to evaluate the best dosage for COQUN ORAL FORMULATION in order to reach a level of plasma concentration which might assure its antioxidant effect if taken on a regular basis.

DETAILED DESCRIPTION:
The study will include 24 healthy subjects who will test the CoQ10 formulation. All 24 subjects will test a single dose of 100mg CoQ10 in 1 day to assess bioavailability, which will be followed by a one week wash-out period and then by a 4 week period of continuous administration of COQUN ORAL FORMULATION in parallel groups (1:1): patients will be divided in the continuous treatment period into two groups, one group of 12 patients with intake of 100mg OD, the other one group of 12 patients with intake of 100mg BID, in order to assess multiple-dose profile of COQUN ORAL FORMULATION.

Patients will have to fast the night before enrolment, for at least 10 hours. Patients will be requested to fill in a short diary in the multidose phase, on a daily basis, for confirming the product correct intake, and informing on any experienced adverse event and eventual medication taken for its solving.

ELIGIBILITY:
Inclusion Criteria:

* Subject Informed consent form (ICF) is signed
* M & F Aged between 35-75 years at the time of the signature of ICF
* A body mass index between 20 and 29 kg/m2
* Fasting the night before enrolment, for at least 10 hours
* Healthy, meaning absence of any prescribed medication for a month prior to the inclusion to the study and during the study
* Willing to avoid a consumption of any food supplements except vitamin D and calcium at least 2 weeks before and during the study
* Consumption of dairy and cereal products (standardized breakfast will include low lactose dairy and bread)
* Willing to follow all study procedures, including attending all site visits (including sessions during which a venous line will be inserted for blood sampling), and keeping a diary for the time of multiple-dose study (to follow their compliance and palatability)

Exclusion Criteria:

* Intake of any prescribed medication within 2 weeks of the beginning of the study
* Intake of any food supplements within 2 weeks of the beginning of the study, except vitamin D and calcium
* Hypotension
* Any clinically significant history of serious digestive tract, liver, kidney, cardiovascular or hematological disease, diabetes
* Gastrointestinal disorders or other serious acute or chronic diseases
* Known lactose/gluten intolerances/ food allergies (limitation for standardization of meals)
* Inadequate veins (in the opinion of the investigator) or known contraindication to placement of a dedicated peripheral line for venous blood withdrawal
* Known drug and/or alcohol abuse
* Using any form of nicotine or tobacco
* Mental incapacity that precludes adequate understanding or cooperation
* Participation in another investigational study or blood donation within 3 months prior to or during this study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Consult Med Iasi, Iași, Iasi County, Romania, Romania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CoQ10 Once Daily: 100 mg OD
  COQUN ORAL FORMULATION: COQUN ORAL FORMULATION is a food supplement based on Coenzyme Q10 MINIACTIVES®
- CoQ10 Twice a Day: 100 mg BID
  COQUN ORAL FORMULATION: COQUN ORAL FORMULATION is a food supplement based on Coenzyme Q10 MINIACTIVES®
Period: Before Randomization
Arm/Group | CoQ10 Once Daily | CoQ10 Twice a Day
Started | 24 | 0
Completed | 24 | 0
Not Completed | 0 | 0
Period: After Randomization
Arm/Group | CoQ10 Once Daily | CoQ10 Twice a Day
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CoQ10 Once Daily | CoQ10 Twice a Day | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (7) | 43 (7) | 39 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Pharmacokinetic Property "Area Under the Curve"
Description: - Area under the curve (microg/ml x h): ≥5
  Due to the explorative aim of the study, descriptive statistics and confidence intervals at 95% level will be provided.
  Data were collected at 1, 2, 4, 8 and 12 hours after intake on the single dose period (day -7) and at each following ambulatory visit.
Time Frame: from day-7 to day 28
Measure: Mean (95% Confidence Interval); unit: microg/l*days
Arm/Group | CoQ10 Once Daily | CoQ10 Twice a Day
Number analyzed (Participants) | 12 | 12
microg/l*days | 2657.45 [2224.3 to 3090.6] | 3459.05 [2806.7 to 4111.4]

2. Primary Outcome: Analysis of Pharmacokinetic Property "Cmax"
Description: - Cmax: ≥0,8
  Due to the explorative aim of the study, descriptive statistics and confidence intervals at 95% level will be provided.
  Data were collected at 1, 2, 4, 8 and 12 hours after intake on the single dose period (day -7) and at each following ambulatory visit.
Time Frame: from day-7 to day 28
Measure: Mean (95% Confidence Interval); unit: microg/l
Arm/Group | CoQ10 Once Daily | CoQ10 Twice a Day
Number analyzed (Participants) | 12 | 12
microg/l | 1163.99 [938.46 to 1389.51] | 1501.89 [1200.32 to 1803.47]

3. Primary Outcome: Analysis of Pharmacokinetic Property "Tmax"
Description: - Tmax: ≥3
  Due to the explorative aim of the study, descriptive statistics and confidence intervals at 95% level will be provided.
  Data were collected at 1, 2, 4, 8 and 12 hours after intake on the single dose period (day -7) and at each following ambulatory visit.
Time Frame: from day-7 to day 28
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | CoQ10 Once Daily | CoQ10 Twice a Day
Number analyzed (Participants) | 12 | 12
hours | 17.5 [11.07 to 23.93] | 16.92 [11.4 to 22.43]

ADVERSE EVENTS:
Time Frame: AE were collected for the total duration of the study (28 days).
Groups:
- CoQ10 Once Daily After Randomization; CoQ10 Once Daily Before Randomization: 100 mg OD
  COQUN ORAL FORMULATION: COQUN ORAL FORMULATION is a food supplement based on Coenzyme Q10 MINIACTIVES®
- CoQ10 Twice a Day After Randomization: 100 mg BID
  COQUN ORAL FORMULATION: COQUN ORAL FORMULATION is a food supplement based on Coenzyme Q10 MINIACTIVES®
Arm/Group | CoQ10 Once Daily After Randomization | CoQ10 Twice a Day After Randomization | CoQ10 Once Daily Before Randomization
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/24
Other Adverse Events (participants affected / at risk) | 0/12 | 3/12 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CoQ10 Once Daily After Randomization (N=12) | CoQ10 Twice a Day After Randomization (N=12) | CoQ10 Once Daily Before Randomization (N=24)
DIZZINESS (Ear and labyrinth disorders) | 0 | 1 | 0
RESPIRATORY VIROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULTACEOUS ANGINA (Cardiac disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03819491/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03819491/SAP_001.pdf